CLINICAL TRIAL: NCT05068752
Title: A Phase II Trial of Vemurafenib in Combination with Sorafenib to Treat Patients with Advanced KRAS Mutated Pancreatic Cancer: Targeting RAF Dimers to Suppress Oncogenic RAS Signaling (The Dr. Nate Nieto Study)
Brief Title: Phase II Trial of Vemurafenib and Sorafenib in Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Bayer (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRI-Vemurafenib-Sorafenib-001
Record Dates: First submitted 2021-09-02; First posted 2021-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreas Cancer
Keywords: Pancreatic cancer; Pancreatic adenocarcinoma; Metastatic; KRAS; Phase 2
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Vemurafenib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vemurafenib in Combination with Sorafenib (Experimental)
  Interventions: Drug: Vemurafenib; Drug: Sorafenib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib 480 mg PO BID daily given with Sorafenib 200 mg PO BID
Drug: Sorafenib — Sorafenib 200 mg PO BID and Vemurafenib 480 mg PO BID daily

SUMMARY:
The purpose of this research is to determine the benefit of two oral chemotherapy drugs, Vemurafenib and Sorafenib, in individuals with KRAS mutated pancreatic cancer who have progressed on standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and be willing to sign the written informed consent for the trial. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Histologically confirmed cancer of the pancreas (KRAS mutated) with metastases and progression on at least ≥ 2 prior treatment regimens for their disease.
4. Known mutation status of KRAS and BRAF kinases. For those patients in which this has not previously been determined, the patient must have an archival tumor specimen (primary or metastatic site) available to submit to confirm KRAS and BRAF status.
5. Have a performance status of 0 or 1 on the ECOG performance scale.
6. Demonstrate adequate organ function
7. Female participants of childbearing potential must have a negative serum pregnancy test performed within 24 hours prior to receiving first dose of trial medication. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
8. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of trial treatment.
9. Male participants must agree to use contraception during the treatment period and for at least 30 days after the last dose of trial treatment and refrain from donating sperm during this period.
10. Patient must have QTC of ≤500ms.
11. Subject must be able to swallow and retain oral medication
12. Measurable disease per RECIST 1.1

Exclusion Criteria:

1. Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent and received trial therapy or used an investigational device within 2 weeks of the first dose of this trials' treatment.
2. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1/Day 1 or who has not recovered (i.e. NCI-CTC AE Version 5.0 ≤ Grade 1 at the time of signing informed consent) from adverse events due to a previously administered agent(s).
3. Previous BRAF inhibitor use such as vemurafenib, GSK2118436 or sorafenib.
4. If patient received major surgery, and has not yet recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Previously untreated or concurrent cancer that is distinct in primary site or histology from pancreatic cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before study entry. All cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form).
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
7. Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v5.0] on repeated measurement) despite optimal medical management.
8. Active of clinically significant cardiac disease
9. Has history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Evidence or history of bleeding diathesis or coagulopathy
12. Patient with any pulmonary hemorrhage/bleeding event of NCI-CTCAE v5.0 ≥ Grade 2 within 4 weeks before initiating study treatment; any other hemorrhage/bleeding event of NCI-CTCAE v5.0 ≥ Grade 3 within 4 weeks before initiating study treatment.
13. Patient with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) within 6 months of informed consent.
14. Presence of a non-healing wound, non-healing ulcer, or bone fracture
15. History of organ allograft (including corneal transplant).
16. Known or suspected allergy or hypersensitivity to any of the study drugs (sorafenib, and or vemurafenib) study drug classes, or excipients of the formulations given during the course of this trial.
17. All patients with known diagnosis of Neurofibromatosis Type 1 or other known RAS-opathies
18. Patients with uncontrolled seizures
19. Treatment with medications that have known risk of QTc interval prolongation or Torsades de Pointe (TdP) within 14 days or 5 half-lives before dose of either drug is given in this study and for the duration of the study. Refer to Appendix E for medications with a known risk of TdP.
20. Treatment with a strong or moderate CYP3A inducers (e.g, phenytoin, carbamazepine, phenobarbital, St. John's Wort [hypericum perforatum], dexamethasone at a dose of greater than 16 mg daily, or rifampin [rifampicin], and/or rifabutin) or inhibitors within 28 days before dose of either drug is given in this study and for the duration of the study. Refer to Appendix G.
21. Malabsorption or other significant bowel or stomach resections
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
23. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
24. Inability to comply with the protocol and/or not willing or not available for follow-up assessments required to assess toxicity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate of Vemurafenib in Combination with Sorafenib | initiation of study treatment until 16 weeks
  To determine the efficacy by the disease control rate (Complete response plus Partial Response plus Stable Disease at 16 weeks) of Vemurafenib in Combination with Sorafenib in patients with KRAS mutated pancreatic cancer.

SECONDARY OUTCOMES:
Confirm the Incidences of Adverse Events of Vemurafenib in Combination with Sorafenib | initiation of study treatment up to 30 days post treatment
  To confirm the incidence of adverse events of Vemurafenib in Combination with Sorafenib in patients with KRAS mutated pancreatic cancer
Clinical Activity of Vemurafenib in Combination with Sorafenib | initiation of study treatment up to study completion, up to 2 years
  To determine the progression free survival of Vemurafenib + Sorafenib in patients with KRAS mutated pancreatic cancer. Progression free survival is defined as first dose treated until the date of progression
Measure circulating ctDNA | initiation of study treatment up to study completion, up to 2 years
  To utilize circulating tumor DNA (ct DNA) in plasma to give qualitative (mutations) and to some extent quantitative (amount of ct DNA) information regarding BRAF and KRAS
Measure phospho ERK and phospho AKT in plasma | initiation of study treatment up to study completion, up to 2 years
  To measure the changes in plasma free DNA in regards to mutated KRAS, phospho ERK and phospho AKT

OTHER OUTCOMES:
Clinical Activity of Vemurafenib in Combination with Sorafenib | initiation of study treatment up to study completion, up to 2 years
  To determine the overall survival of Vemurafenib + Sorafenib in patients with KRAS mutated pancreatic cancer. Overall survival is defined as first dose treated until the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, MS, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No